CLINICAL TRIAL: NCT02825316
Title: Mediterranean Diet vs. Low Residue Diet as an add-on Therapy for Induction of Remission in Patients With Active Crohn's Disease
Brief Title: Mediterranean Diet as an add-on Therapy for Induction of Remission in Patients With Active Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, PhD, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0569-15TLV
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; inflammatory bowel diseases; Mediterranean diet; microbiome
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients with active Crohn's disease that will be allocated to the Mediterranean diet group.
  Interventions: Behavioral: Mediterranean diet
- Group B (Experimental): Patients with active Crohn's disease that will be allocated to the low residue diet group.
  Interventions: Behavioral: Low residue diet

INTERVENTIONS:
Behavioral: Mediterranean diet — Eight weeks course of Mediterranean diet (rich in plant-based food and low in animal protein and fat).
  Arms: Group A
Behavioral: Low residue diet — Eight weeks course of low residue diet (minimal consumption of foods that add residue to the stool, such as raw fruits, vegetables and seeds, as well as nuts, legumes and whole grains).
  Arms: Group B

SUMMARY:
This clinical study is designed to evaluate the effect of Mediterranean diet as an add-on therapy for induction of remission in adult patients with active Crohn's disease and to evaluate its effects on clinical, inflammatory and microbial parameters.

DETAILED DESCRIPTION:
The Mediterranean diet has been associated with anti-inflammatory properties and with decreased risk for several chronic diseases. However, the effect of Mediterranean diet has not been evaluated in patients with inflammatory bowel diseases.

The purpose of this study is to determine whether Mediterranean diet is superior to a low residue diet as an add-on therapy for induction of remission in adult patients with active Crohn's disease and to evaluate its effects on clinical, inflammatory and microbial parameters.

Seventy eligible patients will be randomly assigned to one of two dietary interventions: Mediterranean diet or low residue diet, as an add-on therapy for induction of remission of active Crohn's disease. The effect of the dietary regimens on clinical, inflammatory and microbial parameters will be assessed at 8 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age: 18-75
* Diagnosis of Crohn's Disease
* Montreal classification- B1
* CDAI: 150-450 + CRP>0.5 or fecal calprotectin >200
* Induction therapy with corticosteroids, 5-ASA, AZA, 6-MP, MTX or biologic therapy
* Capacity to give informed consent

Exclusion Criteria:

* Ileostomy or colostomy
* Exclusive enteral nutrition/ partial enteral nutrition
* History of or current severe systemic diseases
* History of admission due to bowel obstruction
* Positive Clostridium difficile toxin
* Positive Salmonella, Shigella, Campylobacter, stool culture
* Pregnancy or lactation
* Use of antibiotics or steroids one month prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) | 8 weeks
  Change from baseline

SECONDARY OUTCOMES:
C-reactive protein | 8 weeks
  Change from baseline
Fecal calprotectin | 8 weeks
  Change from baseline
Remission rate- CDAI<150 + normal CRP/ fecal calprotectin | 52 weeks
Response rate- decrease in 70 points in CDAI + decreased CRP/ fecal calprotectin | 8 weeks
Microbial composition | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Dotan, MD, Principal Investigator — Head, IBD Center, Department of Gastroenterology and Liver Diseases Tel Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No